CLINICAL TRIAL: NCT01661504
Title: Evaluating Violence Against Women Screening in Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Innovations for Poverty Action (Other); Mexican National Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1202009793
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Domestic Violence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Referral Card Only (No Intervention): Women participants at control clinics will be given a referral card containing general information on IPV and a list of resources specific to their community
- Integrated Screening (Experimental): The intervention arm will consist of the following components (described in detail below): a) integrated IPV/Sexual and Reproductive Health Screening, b) supportive care, c) safety planning and harm reduction counseling, d) supported referrals, e) booster counseling sessions at 3 months post-baseline / initial counseling
  Interventions: Behavioral: Integrated Screening

INTERVENTIONS:
Behavioral: Integrated Screening — The intervention arm will consist of the following components (described in detail below): a) integrated IPV/Sexual and Reproductive Health Screening, b) supportive care, c) safety planning and harm reduction counseling, d) supported referrals, e) booster counseling sessions
  Arms: Integrated Screening

SUMMARY:
The overall goal of this proposed study is to develop the state of knowledge in the area of gender-based violence and reproductive health by conducting a randomized controlled trial to improve the health care provider's capacity to screen for intimate partner violence and to mitigate associated risk among women health clinic patrons of reproductive age (ages18-44) with recent experiences of physical or sexual partner violence in Mexico City and its surrounding area.

The specific research objectives are as follows:

1. To increase mid-level health care providers' capacity to identify Intimate Partner Violence (IPV) and assist women with risk mitigation
2. Utilizing a randomized controlled trial, to assess the impact of an enhanced health care worker screening and counselling program on (a) past year severe IPV (sexual or physical), including severe IPV; (b) reproductive coercion (c) use of community-based resources and safety planning; and (d) quality of life; versus minimum standard of care
3. To qualitatively examine which programmatic components may serve as mechanisms for observed changes stated in the second objective
4. To synthesize study findings and a) create recommendations for clinic-based intervention programs to address IPV in low and middle income countries and b) disseminate information as reports, presentation, and peer-reviewed publications

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-44
* Currently in heterosexual relationship with a male partner
* Responds in affirmative to past year sexual or physical violence

Exclusion Criteria:

* Cognitive impairment (slurred speech, inability to follow directions)
* Seeking treatment for life threatening emergency care
* Intends to relocate within 2 years.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 959 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Intimate Partner Violence Victimization from Baseline | 12 months
  Participants will be followed up at 3 months and at 15 months post-baseline to assess intimate partner violence victimization as measured by an adapted Conflict Tactics Scale - 2. This will allow for a 12 month follow-up from the booster counseling session in the intervention group which occurs at 3 months post-baseline.

SECONDARY OUTCOMES:
Change in Quality of Life Score | past month
Change in Use of Community Resources | 12 months
  Adapted Community Resources Checklist
Change in Safety Planning | 12 Months
  Adapted Safety Behavior Checklist
Change in Reproductive Coercion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jhumka Gupta, ScD, Principal Investigator — Yale School of Public Health; Claudia Diaz Olavarrieta, PhD, Principal Investigator — National Institute of Public Health - Mexico; Kathryn L Falb, ScD, Principal Investigator — Yale School of Public Health
Locations (1):
- Health Clinics associated with Ministry of Health in Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Gupta J, Willie TC, Harris C, Campos PA, Falb KL, Garcia Moreno C, Diaz Olavarrieta C, Okechukwu CA. Intimate partner violence against low-income women in Mexico City and associations with work-related disruptions: a latent class analysis using cross-sectional data. J Epidemiol Community Health. 2018 Jul;72(7):605-610. doi: 10.1136/jech-2017-209681. Epub 2018 Mar 7. PMID 29514921
- [Derived] Gupta J, Falb KL, Ponta O, Xuan Z, Campos PA, Gomez AA, Valades J, Carino G, Olavarrieta CD. A nurse-delivered, clinic-based intervention to address intimate partner violence among low-income women in Mexico City: findings from a cluster randomized controlled trial. BMC Med. 2017 Jul 12;15(1):128. doi: 10.1186/s12916-017-0880-y. PMID 28697769
- [Derived] Falb KL, Diaz-Olavarrieta C, Campos PA, Valades J, Cardenas R, Carino G, Gupta J. Evaluating a health care provider delivered intervention to reduce intimate partner violence and mitigate associated health risks: study protocol for a randomized controlled trial in Mexico City. BMC Public Health. 2014 Jul 30;14:772. doi: 10.1186/1471-2458-14-772. PMID 25079882
- See also: protocol paper (published) — http://bmcpublichealth.biomedcentral.com/articles/10.1186/1471-2458-14-772